CLINICAL TRIAL: NCT03121508
Title: Taking on Diabetes to Advance You
Brief Title: Taking on Diabetes to Advance You (TODAY)
Acronym: TODAY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough funding to complete the project as planned
Sponsor: Arlene Schmid (Other)
Responsible Party: Sponsor-Investigator, Arlene Schmid, Associate Professor, Co-Investigator, Colorado State University
Organization: Colorado State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-6245H
Record Dates: First submitted 2017-04-13; First posted 2017-04-20 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The investigators will utilize an evidence-based self-management program, and all individuals will be assigned to the prevention group to promote healthy lifestyles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TODAY Project (Other): All participants will attend individualized self-management sessions led by an occupational therapist. The classes will focus on promoting modifying daily activities, habits, roles, and routines to promote healthy lifestyles for individuals with type 2 diabetes.
  Interventions: Behavioral: Taking on Diabetes to Advance You (TODAY) Project

INTERVENTIONS:
Behavioral: Taking on Diabetes to Advance You (TODAY) Project — This is an individualized educational intervention with activity components designed to assist in modifying habits, roles, and routines to promote healthy lifestyle patterns for individuals with type 2 diabetes.

SUMMARY:
The program will consist of diabetes self-management sessions, led by an occupational therapist. The sessions will be held in an individualized format. Sessions will focus on diabetes education, self-management education, and education on behaviors and adaptive techniques to optimize participation in daily life with type II diabetes. As occupational therapists, the investigators and facilitator, aim to focus on establishing healthy habits, roles, and routines for individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* 18 or older
* patient at the Family Medicine Center in Fort Collins

Exclusion Criteria:

* reading level below 6th grade
* inability to understand written or verbal instructions regarding questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-06-24 (Estimated)

PRIMARY OUTCOMES:
The Diabetes Self-Management Questionnaire | through the end of the intervention period, up to one year
  16-item self-report to assess self-care activities associated with diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Matt Malcolm, PhD, Principal Investigator — Colorado State University
Locations (1):
- Family Medicine Center, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No